CLINICAL TRIAL: NCT00300001
Title: Home-Based Symptom Monitoring: Its Impact on Cancer Care Team Behaviors and Patient Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Community Cancer Care (Other)
Collaborators: Amgen (Industry)
Other Study IDs: 2005-0186
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2006-08-25 (Estimated); Status verified 2006-08

CONDITIONS: Cancer; Solid Tumor; Hematologic Malignancy
Keywords: Cancer; Symptom Management; Supportive Symptom Interventions; Symptom Severity; quality of life; Home-based symptom monitoring
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The primary research objective of this protocol is to evaluate the impact of integrating a home-based symptom monitoring system in the day-to-day care of cancer patients in community settings on the frequency of supportive symptom interventions, symptom severity, and quality of life.

DETAILED DESCRIPTION:
Patients will be randomly assigned to one of two groups. One group will be offered an Internet assisted home-based symptom reporting system Cancer Symptom Monitor (CSM) for a twelve-month study period. Patient and care team evaluations will be measured using quantitative and qualitative methods (via focus groups). The second group will receive "standard care" without home-based symptom monitoring. Both groups will be evaluated at baseline, 1, 2, 3, 6, 9, & 12 months, for symptom levels and overall quality of life during the twelve-month study period.

ELIGIBILITY:
Inclusion Criteria:

18 years old or older Diagnosis of solid tumor or hematologic malignancy Starting active treatment (chemotherapy or hormonal therapy) Must be able to give informed consent & consent to use the Cancer Symptom Monitor -

Exclusion Criteria:

Inability to give informed consent Life expectancy of less than 3 months Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Dale E. Theobald, PhD, MD, Principal Investigator — Community Cancer Care, Inc.
Locations (3):
- United States (3):
  - Quality Oncology Care, Inc., Indianapolis, Indiana
  - Community Regional Cancer Center-Community Hospital North, Indianapolis, Indiana
  - Morgan Hospital and Medical Center, Martinsville, Indiana

REFERENCES:
- [Background] Berger AM, Portenoy RK, Weissman DE., Eds. Principles and Practice of Supportive Oncology, 2nd Ed.; Lippincott-Raven: Philadelphia, 2002.
- [Background] Max MB, Portenoy RK, Laska EM, Eds. Oxford Textbook of Palliative Medicine, 2nd Ed.; Oxford Medical Publications: New York, 1998.
- [Background] Cleeland CS, Reyes-Gibby CC. When is it justified to treat symptoms? Measuring symptom burden. Oncology (Williston Park). 2002 Sep;16(9 Suppl 10):64-70. PMID 12380956
- [Background] Chang VT, Ingham J. Symptom control. Cancer Invest. 2003;21(4):564-78. doi: 10.1081/cnv-120022376. PMID 14533447
- [Background] Patrick DL, Ferketich SL, Frame PS, Harris JJ, Hendricks CB, Levin B, Link MP, Lustig C, McLaughlin J, Ried LD, Turrisi AT 3rd, Unutzer J, Vernon SW; National Institutes of Health State-of-the-Science Panel. National Institutes of Health State-of-the-Science Conference Statement: Symptom Management in Cancer: Pain, Depression, and Fatigue, July 15-17, 2002. J Natl Cancer Inst. 2003 Aug 6;95(15):1110-7. doi: 10.1093/jnci/djg014. PMID 12902440
- [Background] Oncology Nursing Society, Research Agenda, 2003-2205. Available at http://www.ons.org/images/PDFs/Research/2003Plan.pdf.
- [Background] Passik SD, Dugan W, McDonald MV, Rosenfeld B, Theobald DE, Edgerton S. Oncologists' recognition of depression in their patients with cancer. J Clin Oncol. 1998 Apr;16(4):1594-600. doi: 10.1200/JCO.1998.16.4.1594. PMID 9552071
- [Background] McDonald MV, Passik SD, Dugan W, Rosenfeld B, Theobald DE, Edgerton S. Nurses' recognition of depression in their patients with cancer. Oncol Nurs Forum. 1999 Apr;26(3):593-9. PMID 10214600
- [Background] Abdullah M, Theobald DE, Butler D, Kroenke K, Perkins A, Edgerton S, Dugan WM Jr. Access to communication technologies in a sample of cancer patients: an urban and rural survey. BMC Cancer. 2005 Feb 17;5:18. doi: 10.1186/1471-2407-5-18. PMID 15717933
- [Background] Theobald DE, Butler D, Coburn J, et al. IVR-based cancer symptom assessment: Nurses' expectations and perceived barriers. (Abstract) Am Soc Clin Oncol, New Orleans, 2004.
- [Background] Sonis ST, Elting LS, Keefe D, Peterson DE, Schubert M, Hauer-Jensen M, Bekele BN, Raber-Durlacher J, Donnelly JP, Rubenstein EB; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Perspectives on cancer therapy-induced mucosal injury: pathogenesis, measurement, epidemiology, and consequences for patients. Cancer. 2004 May 1;100(9 Suppl):1995-2025. doi: 10.1002/cncr.20162. PMID 15108222
- [Background] Cleeland CS, Mendoza TR, Wang XS, Chou C, Harle MT, Morrissey M, Engstrom MC. Assessing symptom distress in cancer patients: the M.D. Anderson Symptom Inventory. Cancer. 2000 Oct 1;89(7):1634-46. doi: 10.1002/1097-0142(20001001)89:73.0.co;2-v. PMID 11013380
- [Background] Schubert MM, Williams BE, Lloid ME, Donaldson G, Chapko MK. Clinical assessment scale for the rating of oral mucosal changes associated with bone marrow transplantation. Development of an oral mucositis index. Cancer. 1992 May 15;69(10):2469-77. doi: 10.1002/1097-0142(19920515)69:103.0.co;2-w. PMID 1568168
- [Background] Kreuger RA. Focus Groups: A practical guide for Applied Research. Sage Publications: Thousand Oakes, CA, 1994.
- [Background] Munhall P. Nursing Research: A qualitative perspective, third edition. 2001.
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Morgan, D. Focus Groups as Qualitative Research. Sage Publications. Thousand Oakes, CA, 1997.